CLINICAL TRIAL: NCT02748109
Title: Assessment and Rehabilitation of Central Sensory Impairments for Balance in mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie King, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15010; CDMRP-MR141257 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2016-03-29; First posted 2016-04-22 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Brain Injury
Keywords: Physical Therapy; Balance Disorder; Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vestibular Rehabilitation + audio biofeedback (Experimental): Vestibular rehabilitation paired with audio biofeedback
  Interventions: Behavioral: Vestibular Rehabilitation + audio biofeedback
- Vestibular Rehabilitation (Active Comparator): Vestibular rehabilitation
  Interventions: Behavioral: Vestibular Rehabilitation

INTERVENTIONS:
Behavioral: Vestibular Rehabilitation + audio biofeedback — Vestibular rehabilitation paired with audio biofeedback for balance control 2 times per week with a physical therapist for 6 weeks.
  Arms: Vestibular Rehabilitation + audio biofeedback
Behavioral: Vestibular Rehabilitation — Standard vestibular rehabilitation 2 times per week with a physical therapist for 6 weeks.
  Arms: Vestibular Rehabilitation

SUMMARY:
Our central hypothesis is that chronic balance deficits after mild traumatic brain injury (mTBI) result from impairments in central sensorimotor integration (CSMI) that may be helped by rehabilitation. There are two objectives of this proposal; the first objective is to characterize balance deficits in people with mTBI. The second objective is to use a novel auditory bio-feedback (ABF) device to improve measures central sensorimotor integration and balance control.

DETAILED DESCRIPTION:
Objectives: This study as two parts: 1) Cross-sectional study (Aim I: Balance Assessment) to identify and characterize maladaptive balance control strategies after mTBI compared to healthy controls and 2) Interventional randomized pilot study (Aim II: Balance Rehabilitation) using a novel ABF rehabilitation technique to ameliorate maladaptive balance control strategies after TBI. Subjects in Aim II will be a subset from Aim I and studies will occur simultaneously.

Plan: The proposed 4-year study has two parts: 1) Cross-sectional study (Aim I: Balance Assessment) to identify and characterize maladaptive balance control strategies after mTBI compared to healthy controls and 2) Interventional randomized pilot study (Aim II: Balance Rehabilitation) using a novel ABF rehabilitation technique to ameliorate maladaptive balance control strategies after TBI. Subjects in Aim II will be a subset from Aim I and studies will occur simultaneously.

Methods: I) Balance Assessment: To characterize balance deficits in people with mTBI who have chronic, non-resolving balance deficits compared to healthy control subjects without a history of mTBI. We hypothesize that a) objective measures of central sensorimotor integration, static and dynamic balance will better distinguish people with mTBI from control subjects than clinical measures, b) a subset of people with mTBI will have abnormal central sensori-motor integration (CSMI) test measures, even without peripheral vestibular or ocular motor deficits c) the relationship between poorer static/dynamic balance performance and mTBI is regulated/mediated by CSMI. We will test 130 subjects between the ages of 18 and 60; 65 with chronic (> 3 months) mTBI and non-resolving balance deficits and 65 healthy age and gender matched control subjects without a history of mTBI. We will obtain objective measures of static and dynamic balance using wearable inertial sensors and determine how these measures relate to central sensorimotor integration. We will also obtain laboratory measures of peripheral vestibular function and ocular motor function to help classify people and to consider as potential covariates in rehabilitation efficacy.

II) Balance Rehabilitation: To determine the efficacy of a novel, ABF balance rehabilitation program to improve central sensorimotor integration, static and dynamic balance, and functional activity in patients with chronic mTBI. We hypothesize that a) CSMI scores will improve with rehabilitation and ABF will increase the improvement of CSMI scores beyond the standard of care, b) ABF intervention will improve objective summary measures of balance and c) people with central sensorimotor integration impairment will show sustained improvement in CSMI scores and balance after rehabilitation. We will randomize 40 subjects between the ages of 18 and 60; 65 with chronic (> 3 months) mTBI and non-resolving balance deficits from Aim I who have abnormal CSMI into either the ABF rehabilitation group or the standard of care group. People will be tested before and after a 6-week intervention period and again 6 week later to determine long-term changes. Normal/abnormal vestibular and ocular motor function will be used as covariates to determine if peripheral deficits affect the efficacy of ABF rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of mTBI based upon Veterans Health Administration (VHA)/Department of Defense (DoD) criteria with persisting symptoms >3 months post injury
* have minimal cognitive impairment; a score between 0 and 8 on the Short Blessed test for cognitive function
* may have or not had a loss of consciousness (LOC) with their initial injury

-OR-

* have no recent history of mTBI or brain injury and related complaints

Exclusion Criteria:

* have had or currently have any other injury, medical, substance or neurological illness that could potentially explain balance deficits (e.g., Central Nervous System disease, stroke, moderate TBI, lower extremity amputation)
* meet criteria for moderate to severe substance use disorder within the past month, as defined by Diagnostic and Statistical Manual (DSM-V)
* display behavior that would significantly interfere with validity of data collection or safety during study
* be in significant pain during the evaluation (5/10 by patient subjective report)
* be a pregnant female (balance considerations)
* have past history of peripheral vestibular pathology or ocular motor deficits
* have significant hearing loss that would interfere with the use of an auditory biofeedback device; hearing loss no worse than 30 decibel (dB) HL (PTA 0.5-3 kHz), in better ear, with the difference in ears being less than 15 dB PTA
* be unable to abstain for 24 hours in advance of testing in the use medications that might impair their balance (meclizine, scopolamine, benzodiazepines such as Valium, sedatives such as Ambien, narcotic pain medications, and antihistamines)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Change in gait activity in the home as measured using an inertial sensor continuously in the home for a week before and after intervention. | before and after 6 weeks of intervention
  An APDM movement monitor will be worn around the waist to gather information on local activity during the day.

SECONDARY OUTCOMES:
Change in Sensory Orientation Test (SOT) Composite Score | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare baseline SOT composite score with the post rehabilitation scores looking for a difference between the standard of care and audio biofeedback rehabilitation groups.
Change in Modified Balance Error Scoring System (mBESS) instrumented and non-instrumented scores | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare baseline mBESS measures using inertial sensors and the clinical scoring method looking for a difference between the standard of care and audio biofeedback rehabilitation groups.
Change in dynamic gait coordination | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare baseline gait measures using inertial sensors looking for a difference between the standard of care and audio biofeedback rehabilitation groups.
Change in Sport Concussion Assessment Tool - 3rd edition (SCAT-3) symptoms questionnaire | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare subjects symptoms using the SCAT-3 symptom log looking for a difference between the standard of care and audio biofeedback rehabilitation groups.
Automated Neuropsychological Assessment Metrics (ANAM) | baseline
  We will use this test to determine if it is a good predictor for rehabilitation outcomes
Dizziness Handicap Index (DHI) | baseline
  This questionnaire takes approximately 10 minutes and asks if you become dizzy while performing various tasks.
PTSD Checklist | baseline
  This questionnaire takes approximately 10 minutes and is a list of problems and complaints some people have in response to stressful life experiences.
Pain Location Inventory | baseline
  This questionnaire takes approximately 5 minutes and asks if you have pain and where that pain is located.
SIQR symptom Questionnaire | baseline
  This questionnaire asks you to rate different symptoms on a sliding scale.
Sports Concussion Assessment Tool - 3 (SCAT-3) symptom questionnaire | Every session
  This questionnaire takes approximately 5 minutes and asks you to rate 22 different symptoms on a scale between zero and six.
Becks Depression Inventory (BDI) | baseline
  This questionnaire takes approximately 5 minutes and will ask questions regarding depression and personal emotions.
Short Form - 36 | baseline
  This questionnaire will take approximately 10 minutes and covers 36 questions about daily living and how your symptoms have or have not changed over certain time periods.
Neurobehavioral Symptom Inventory | baseline
  This questionnaire takes approximately 10 minutes and goes through commons symptoms after traumatic brain injury (such as nausea and blurred vision) and asks you to rate your symptoms.
Change in Central Sensorimotor Integration (CSMI) Weighting Scores; vision | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare baseline CSMI scores (Wvis) with post rehabilitation scores looking for a difference between the standard of care and audio biofeedback rehabilitation groups.
Change in Central Sensorimotor Integration (CSMI) Weighting Scores; vestibular | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare baseline CSMI scores (Wvest) with post rehabilitation scores looking for a difference between the standard of care and audio biofeedback rehabilitation groups.
Change in Central Sensorimotor Integration (CSMI) Weighting Scores; proprioception | Subjects will be tested before and after a 6-week intervention period and again 6 weeks later to determine long-term changes
  We will compare baseline CSMI scores (Wprop) with post rehabilitation scores looking for a difference between the standard of care and audio biofeedback rehabilitation groups.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie King, Ph.D., P.T., Principal Investigator — Associate Professor of Neurology, OHSU
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fino PC, Raffegeau TE, Parrington L, Peterka RJ, King LA. Head stabilization during standing in people with persisting symptoms after mild traumatic brain injury. J Biomech. 2020 Nov 9;112:110045. doi: 10.1016/j.jbiomech.2020.110045. Epub 2020 Sep 17. PMID 33011672
- [Background] Stuart S, Parrington L, Morris R, Martini DN, Fino PC, King LA. Gait measurement in chronic mild traumatic brain injury: A model approach. Hum Mov Sci. 2020 Feb;69:102557. doi: 10.1016/j.humov.2019.102557. Epub 2019 Nov 26. PMID 31783306
- [Background] Martini DN, Parrington L, Stuart S, Fino PC, King LA. Gait Performance in People with Symptomatic, Chronic Mild Traumatic Brain Injury. J Neurotrauma. 2021 Jan 15;38(2):218-224. doi: 10.1089/neu.2020.6986. Epub 2020 Aug 10. PMID 32495691
- [Background] Stuart S, Parrington L, Martini DN, Kreter N, Chesnutt JC, Fino PC, King LA. Analysis of Free-Living Mobility in People with Mild Traumatic Brain Injury and Healthy Controls: Quality over Quantity. J Neurotrauma. 2020 Jan 1;37(1):139-145. doi: 10.1089/neu.2019.6450. Epub 2019 Aug 26. PMID 31354032
- [Background] Peterka RJ, Murchison CF, Parrington L, Fino PC, King LA. Implementation of a Central Sensorimotor Integration Test for Characterization of Human Balance Control During Stance. Front Neurol. 2018 Dec 13;9:1045. doi: 10.3389/fneur.2018.01045. eCollection 2018. PMID 30619027
- [Background] Fino PC, Wilhelm J, Parrington L, Stuart S, Chesnutt JC, King LA. Inertial Sensors Reveal Subtle Motor Deficits When Walking With Horizontal Head Turns After Concussion. J Head Trauma Rehabil. 2019 Mar/Apr;34(2):E74-E81. doi: 10.1097/HTR.0000000000000418. PMID 30045224
- [Background] Fino PC, Parrington L, Walls M, Sippel E, Hullar TE, Chesnutt JC, King LA. Abnormal Turning and Its Association with Self-Reported Symptoms in Chronic Mild Traumatic Brain Injury. J Neurotrauma. 2018 May 15;35(10):1167-1177. doi: 10.1089/neu.2017.5231. Epub 2018 Mar 23. PMID 29078732
- [Background] Fino PC, Peterka RJ, Hullar TE, Murchison C, Horak FB, Chesnutt JC, King LA. Assessment and rehabilitation of central sensory impairments for balance in mTBI using auditory biofeedback: a randomized clinical trial. BMC Neurol. 2017 Feb 23;17(1):41. doi: 10.1186/s12883-017-0812-7. PMID 28231824
- [Background] Theodoroff SM, Papesh M, Duffield T, Novak M, Gallun F, King L, Chesnutt J, Rockwood R, Palandri M, Hullar T. Concussion Management Guidelines Neglect Auditory Symptoms. Clin J Sport Med. 2022 Mar 1;32(2):82-85. doi: 10.1097/JSM.0000000000000874. PMID 32941367